CLINICAL TRIAL: NCT02961101
Title: Anti-PD-1 Antibody Alone or in Combination With Low-dose Decitabine and/or Chemotherapy in Relapsed or Refractory Malignancies: an Open-label Phase I/II Trial
Brief Title: Anti-PD-1 Antibody Alone or in Combination With Decitabine/Chemotherapy in Relapsed or Refractory Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Han weidong (Other)
Responsible Party: Sponsor-Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-019
Record Dates: First submitted 2016-11-02; First posted 2016-11-10 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Malignancies Multiple
Keywords: relapsed or refractory; malignancies; decitabine; anti-PD-1 antibody; chemotherapy
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — spartalizumab; Decitabine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anti-PD-1 antibody+decitabine (Experimental): Decitabine will be administrated at 10mg/d on day1 to 5, followed by Anti-PD-1 antibody 200mg on day8 IV Q3 weeks until progression.
  Interventions: Drug: Anti-PD-1 antibody; Drug: Decitabine
- Anti-PD-1 antibody (Experimental): Anti-PD-1 antibody 200mg IV Q3 weeks until progression.
  Interventions: Drug: Anti-PD-1 antibody
- Anti-PD-1 antibody+chemotherapy (Experimental): Chemotherapy will be given depends on the cancer type and treatment regimen before enrollment. Chemotherapy was administrated on day1 , followed by Anti-PD-1 antibody 200mg on day2 IV Q3 weeks until progression. Following disease remission, radiotherapy could be administered or omitted for consolidation at the discretion of the investigator.
  Interventions: Drug: Anti-PD-1 antibody; Drug: Chemotherapy

INTERVENTIONS:
Drug: Anti-PD-1 antibody — Anti-PD-1 antibody will be given at 1-3mg/kg on day8 by IV every three weeks
Drug: Decitabine — Decitabine will be given at 10mg/d on day 1to 5 by IV every three weeks
  Arms: Anti-PD-1 antibody+decitabine
Drug: Chemotherapy — Chemotherapy be given depends on the cancer type and treatment regimen before enrollment.
  Arms: Anti-PD-1 antibody+chemotherapy

SUMMARY:
The purpose of this study is to assess the feasibility, safety, and efficacy of anti-PD-1 antibody alone or in combination with low-dose decitabine in patients with relapsed or refractory malignancies, including Non-Hodgkin'lymphoma, Hodgkin'lymphoma, gastrointestinal cancers, hepatocellular carcinoma, breast cancer, ovarian cancer or lung cancer or renal-cell cancer or pancreatic cancer or bile duct cancer.

DETAILED DESCRIPTION:
Primary objective: To assess the feasibility and safety for Anti-PD-1 antibody alone or in combination with decitabine and/or chemotherapy administered every 3 weeks to subjects with relapsed or refractory malignancies.

Secondary objectives: 1) To assess the antitumor activity of Anti-PD-1 antibody alone or in combination with decitabine and/or chemotherapy in subjects with relapsed or refractory malignancies. 2) To characterize the immunological effects of Anti-PD-1 antibody alone or in combination with decitabine and/or chemotherapy. 3) To characterize the immunological effects of Anti-PD-1 antibody alone or in combination with decitabine and/or chemotherapy.

Exploratory objectives: 1) To analysis of potential biological parameters correlated to clinical response and toxicities. 2) To search predictive biomarkers to guide the choose of patients undergoing the treatment of Anti-PD-1 antibody alone or in combination with decitabine and/or chemotherapy.

Safety Evaluation: Adverse events will be assessed continuously during the study and for 100 days post last treatment, and will be evaluated according to the NCI CTCAE Version 4.0.

Efficacy Evaluation: 1) Treatment response to lymphoma was defined using the International Workshop to Standardize Response Criteria for Lymphomas; 2) Treatment response to solid tumors was defined using Response Evaluation Criteria in Solid Tumors (RECIST1.1).

evaluation index: BOR; ORR; PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological confirmation of relapsed or refractory malignancies,including Non-Hodgkin'lymphoma, Hodgkin'lymphoma, gastrointestinal cancers, hepatocellular carcinoma, breast cancer, ovarian cancer or lung cancer or renal-cell cancer or pancreatic cancer or bile duct cancer.
2. 12 to 75 years of age.
3. ECOG performance of less than 2.
4. Life expectancy of at least 3 months.
5. Subjects with lymphoma must have at least one measureable lesion >1 cm as defined by lymphoma response criteria; with solid tumors must have at least one measureable lesion >1 cm per RECIST1.1.
6. Subjects must have received at least two prior chemotherapy regimen, and must be off therapy for at least 4 weeks prior to Day 1. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months.
7. Subjects must have adequate bone marrow, live, renal, lung and heart functions.

   1. Absolute neutrophil count greater than or equal to 1,000/μL.
   2. Platelet count greater than or equal to 70,000/µL.
   3. Serum bilirubin level less than or equal to 1.5 x upper limits of normal (ULN).
   4. Serum creatinine less than or equal to 1.5 x ULN.
   5. Alanine aminotransferase [ALT or SGPT] and aspartate aminotransferase [AST or SGOT] less than or equal to 2.5 x ULN.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary and intestinal infection especially.
3. Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in 1 month .
4. Prior organ allograft.
5. Women who are pregnant or breastfeeding.
6. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 2 years

SECONDARY OUTCOMES:
Objective response by Response Evaluation Criteria in Solid Tumors (RECIST1.1). | 3 years
Objective response by the International Workshop to Standardize Response Criteria for lymphomas. | 3 years
Progression free survival | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Chunmeng Wang, Master, Study Director — Biotherapeutic Department of Chinese PLA General Hospital, Beijing, China, 100853; Wenying Zhang, Master, Study Director — Biotherapeutic Department of Chinese PLA General Hospital, Beijing, China, 100853; Yang Liu, Doctor, Study Director — Biotherapeutic Department of Chinese PLA General Hospital, Beijing, China, 100853; Meixia Chen, Doctor, Study Director — Biotherapeutic Department of Chinese PLA General Hospital, Beijing, China, 100853; Yan Zhang, Doctor, Principal Investigator — Biotherapeutic Department of Chinese PLA General Hospital, Beijing, China, 100853; Qian Mei, Doctor, Study Director — Department of Molecular Biology, Institute of Basic Medicine, Chinese PLA General Hospital, Beijing, 100853, China.; Jing Nie, Doctor, Study Director — Department of Molecular Biology, Institute of Basic Medicine, Chinese PLA General Hospital, Beijing, 100853, China.; Xiang Li, Master, Principal Investigator — Department of Molecular Biology, Institute of Basic Medicine, Chinese PLA General Hospital, Beijing, 100853, China.; Liang Dong, Master, Principal Investigator — Department of Molecular Biology, Institute of Basic Medicine, Chinese PLA General Hospital, Beijing, 100853, China.; Lu Shi, Master, Principal Investigator — Department of Molecular Biology, Institute of Basic Medicine, Chinese PLA General Hospital, Beijing, 100853, China.; Kaichao Feng, Doctor, Principal Investigator — Biotherapeutic Department of Chinese PLA General Hospital, Beijing, China, 100853; Jingdan Qiu, Doctor, Principal Investigator — Biotherapeutic Department of Chinese PLA General Hospital, Beijing, China, 100853; Hejin Jia, Doctor, Principal Investigator — Biotherapeutic Department of Chinese PLA General Hospital, Beijing, China, 100853
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Mei Q, Chen M, Lu X, Li X, Duan F, Wang M, Luo G, Han W. An open-label, single-arm, phase I/II study of lower-dose decitabine based therapy in patients with advanced hepatocellular carcinoma. Oncotarget. 2015 Jun 30;6(18):16698-711. doi: 10.18632/oncotarget.3677. PMID 25895027
- [Result] Nie J, Zhang Y, Li X, Chen M, Liu C, Han W. DNA demethylating agent decitabine broadens the peripheral T cell receptor repertoire. Oncotarget. 2016 Jun 21;7(25):37882-37892. doi: 10.18632/oncotarget.9352. PMID 27191266
- [Derived] Liu Y, Wang C, Li X, Dong L, Yang Q, Chen M, Shi F, Brock M, Liu M, Mei Q, Liu J, Nie J, Han W. Improved clinical outcome in a randomized phase II study of anti-PD-1 camrelizumab plus decitabine in relapsed/refractory Hodgkin lymphoma. J Immunother Cancer. 2021 Apr;9(4):e002347. doi: 10.1136/jitc-2021-002347. PMID 33820822
- [Derived] Wang C, Liu Y, Dong L, Li X, Yang Q, Brock MV, Mei Q, Liu J, Chen M, Shi F, Liu M, Nie J, Han W. Efficacy of Decitabine plus Anti-PD-1 Camrelizumab in Patients with Hodgkin Lymphoma Who Progressed or Relapsed after PD-1 Blockade Monotherapy. Clin Cancer Res. 2021 May 15;27(10):2782-2791. doi: 10.1158/1078-0432.CCR-21-0133. Epub 2021 Mar 5. PMID 33674274
- [Derived] Nie J, Wang C, Liu Y, Yang Q, Mei Q, Dong L, Li X, Liu J, Ku W, Zhang Y, Chen M, An X, Shi L, Brock MV, Bai J, Han W. Addition of Low-Dose Decitabine to Anti-PD-1 Antibody Camrelizumab in Relapsed/Refractory Classical Hodgkin Lymphoma. J Clin Oncol. 2019 Jun 10;37(17):1479-1489. doi: 10.1200/JCO.18.02151. Epub 2019 Apr 30. PMID 31039052